CLINICAL TRIAL: NCT05291494
Title: A Study on the Effectiveness of WeChat-based Online Education to Reduce Perioperative Anxiety in Breast Cancer Patients: a Prospective Randomized Controlled Study
Brief Title: A Study on the Effectiveness of WeChat-based Online Education to Reduce Perioperative Anxiety in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-1138
Record Dates: First submitted 2021-12-29; First posted 2022-03-22 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer Female
Keywords: periperative anxiety

STUDY DESIGN:
Intervention Model Description: The experimental group will watch science videos through WeChat and regular preoperative visits before the surgical procedures. The regular group only received regular preoperative visits and education by ward nurses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, the anesthesiologist, data collectors, the physicians performing the follow-up, and data analysts will be blinded to the group allocation. Blinding will maintain until the completion of the final analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WeChat group (Experimental): The patients in this group will be first assessed by a researcher on admission about anxiety and sleep (base on the State-Trait Anxiety Inventory (STAI) scale and the sleep quality scale (SQS)). Once the assessment completed, the patients are required to follow the WeChat public platform to watch the education videos when they are free. The content of the videos covers all aspects of surgery, anesthesia, and perioperative care. The videos are presented in an easy-to-understand pattern to ensure participants of all ages and levels of education comfortably understand the content.
  Interventions: Behavioral: follow the WeChat public platform to watch the education videos
- Regular group (Placebo Comparator): Patients in this group were also assessed by the same researcher on admission for anxiety and sleep (base on State-Trait Anxiety Inventory (STAI) scale; sleep quality scale (SQS) scale). Upon completion of the assessment, they received oral instruction from the ward nurse covering the same contents as above instead of the education video.
  Interventions: Behavioral: regular preoperative visits and education by ward nurses.

INTERVENTIONS:
Behavioral: follow the WeChat public platform to watch the education videos — In addition to the regular preoperative visits, the WeChat education group will watch science videos through WeChat before the surgical procedures.
  Arms: WeChat group
Behavioral: regular preoperative visits and education by ward nurses. — received oral instruction from the ward nurse covering the same contents as above instead of the education video.
  Arms: Regular group

SUMMARY:
Patients who meet the enrollment criteria will be randomly assigned to the WeChat education group and the regular group. In addition to the regular preoperative visits, the WeChat education group will also watch science videos through WeChat before the surgical procedures. The regular group only received regular preoperative visits and education by ward nurses. The main observation indicator is the incidence of preoperative anxiety defined as the scores of State Anxiety Inventory more than 40 points.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will be randomly assigned to the WeChat online education group or the regular group. Two researchers will conduct preoperative education, preoperative evaluation and postoperative follow-up respectively.The patients in WeChat group will be first assessed by a researcher on admission about anxiety and sleep (base on the State-Trait Anxiety Inventory (STAI) scale and the sleep quality scale (SQS)). Once the assessment completed, the patients are required to follow the WeChat public platform to watch the education videos when they are free. The content of the videos is jointly decided by the breast surgeon, anesthetists, and ward nurse including the overall prognosis, surgical approach, postoperative rehabilitation exercises, preparation for anesthesia, anesthesia approach and possible effects of anesthesia, which covers all aspects of surgery, anesthesia, and perioperative care. The videos are presented in an easy-to-understand pattern to ensure participants of all ages and levels of education comfortably understand the content. Participants can simply click on the video dialogue box in the public platform for playback and watch it unconditionally.Patients in regular group will be also assessed by the same researcher on admission for anxiety and sleep (base on State-Trait Anxiety Inventory (STAI) scale; sleep quality scale (SQS) scale). Upon completion of the assessment, they received oral instruction from the ward nurse covering the same contents as above instead of the education video.

ELIGIBILITY:
Inclusion Criteria:

* female patients scheduled for elective breast cancer resection;
* aged 18 to 80 years,;
* American Society of Anesthesiologists (ASA) physical status I-III.

Exclusion Criteria:

* patients diagnosed with primary breast cancer combined with malignant tumors of other organs (such as lung, kidney, intestine, etc.);
* patients with tumor recurrence after reoperation;
* patients failing to cooperate with the study for any reason, such as communication disorders.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
the incidence of preoperative anxiety | The day before surgery
  The primary outcome indicator is the incidence of preoperative anxiety, defined as a S-AI(The State Anxiety Inventory)score of >40.The total S-AI score ranges from 20 to 80, with higher scores indicating more severe anxiety.When S-AI score exceeds 40, a state of clinical anxiety is confirmed25,26.A S-AI score outstripping 44 strongly denotes severe anxiety.

SECONDARY OUTCOMES:
incidence of severe anxiety (S-AI > 44) on 1day before and at 72 hours after surgery | The day before and at 72 hours after surgery
  Subjects will be assessed for anxiety on 1day before and at 72 hours after surgery
incidence of anxiety 72 hours after surgery | at 72 hours after surgery
  Subjects will be assessed for anxiety on 1day before and at 72 hours after surgery
NRS scores for pain at rest and during movement | at 24，48 , 72 hours after surgery
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
incidence of PONV within 24 hours after surgery | during the first 24 hours after surgery
  the investigators considered it PONV if patients felt any nausea or had any vomiting
subjective sleep score (Sleep Quality Score (SQS)) | At 1 week after surgery
  subjective sleep score(Sleep Quality Score (SQS)) at 1 week postoperatively.SQS is a self-assessment questionnaire with discrete visual analog scale (VAS). The questionnaire asked the respondents to score the overall sleep quality of the 7-day recall period on a discrete VAS scale. The respondents scored on the following five categories, with a score of 0 to 10:0 = bad, 1-3 = poor, 4-6 = fair, 7-9 = good and 10 = very good.
quality of life QoR-15 scores at 1 and 3 months postoperatively | at 1 and 3 months after surgery
  The investigators use the 15-item quality of recovery score (QoR-15 questionnaire) to reveal the life quality.QoR-15 consists of 15 questionnaires to assess patients' postoperative recovery, each of which is based on the pain rating scale and constructs an 11-point numerical rating scale. For positive items, 0 = never and 10 = always; For negative items, the score was reversed, and the final score was the sum of the 15 items, with the highest score being 150. The higher the score, the better the postoperative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao X, Zuo YD, Kuang SY, Liu CY, Kun-Shao, Wang H, Yan SY, Yu F, Xu Y, Zhou L, Jiang CL. Effectiveness of WeChat-assisted preoperative education to reduce perioperative anxiety in breast cancer patients: a prospective randomized controlled study protocol. Trials. 2024 Apr 3;25(1):231. doi: 10.1186/s13063-024-08071-3. PMID 38570855